CLINICAL TRIAL: NCT00725400
Title: Phase II Open Label Comparative Study of Cetuximab and Radiation Therapy Vs Surgery Before or After Radiation Therapy in Patients With Stage II to IV Colorectal Carcinoma
Brief Title: Comparative Study of Cetuximab and Radiation Vs Surgery Before or After Radiation in Patients With Colorectal Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn due to unavailability of eligible subject population. We will request the sponsors to extend the time for enrollment.
Sponsor: American Scitech International (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Dr. Ratna Grewal, American Scitech International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-CRO0000192008; JLRH-0000292008; IORG-0000392008; BMS-192008; IMCL-II-ASI-IORG-92008; ASI-CRCII0708
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Colorectal Carcinoma
Keywords: Colorectal Cancer; Erbitux; Cetuximab; Surgery; Radiation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will receive a Cetuximab and Radiation Therapy.
  Interventions: Other: Cetuximab and Radiation Therapy
- 2 (Active Comparator): Patients will undergo Surgery before or after Radiation Therapy.
  Interventions: Procedure: Surgery and Radiation Therapy

INTERVENTIONS:
Other: Cetuximab and Radiation Therapy — Patients will receive Cetuximab and Radiation Therapy. Patients will receive a dose of Cetuximab through Intravenous (IV). The initial dose is 400 mg/m2 administered as a 120-minute intravenous infusion (maximum infusion rate 10 mg/min) and weekly dose is 250 mg/m2 infused over 60 minutes (maximum infusion rate 10 mg/min) until disease progression or unacceptable toxicity. Radiation treatment for Colorectal Cancer are Intensity Modulated Radiation Therapy (IMRT). IMRT delivers radiation directly to the tumor and modulates the intensity of the radiation with laser accuracy.
  Other Names: Erbitux and Radiotherapy
  Arms: 1
Procedure: Surgery and Radiation Therapy — Patients will undergo Surgery before or after Radiation Therapy. Colorectal Cancer Surgery are Colon resection (Colectomy), Rectum resection (Proctectomy), Colostomy, and Radiofrequency ablation. Radiation treatment for Colorectal Cancer are Intensity Modulated Radiation Therapy (IMRT). IMRT delivers radiation directly to the tumor and modulates the intensity of the radiation with laser accuracy.
  Other Names: Surgery and Radiotherapy
  Arms: 2

SUMMARY:
RATIONALE: Monoclonal antibodies, such as Cetuximab, can target tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.This is an anti-cancer drug which has already been approved by the FDA for use in patients who have Colorectal Cancer. Cetuximab can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation Therapy uses high-energy x-rays to kill tumor cells and cause less damage to normal tissue . Giving the drug Cetuximab together with Radiation Therapy may kill more tumor cells. Surgery is the most common treatment for Colorectal Cancer to remove the tumor, as well as a small margin of surrounding normal tissue and possibly nearby lymph nodes. Surgery is usually used in conjunction with other conventional treatments such as Radiation Therapy. Radiation Therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation Therapy after surgery may kill any tumor cells that remain after surgery.

Screening test such as Fecal Occult Blood Test (FOBT) and Colonoscopy has to be done. Tumor markers for Colorectal Carcinoma are Carcinoembryonic antigen (CAE) and CA 19-9 and to assess the response of tumor markers Carcinoembryonic antigen (CAE) and CA 19-9 will be used and periodically Colonoscopy has to be done. Colorectal Cancer Surgery are Colon resection (Colectomy), Rectum resection (Proctectomy), Colostomy, and Radiofrequency ablation.

PURPOSE: Determine the tumor response rate treated with Cetuximab and Radiation Therapy Vs Surgery before or after Radiation Therapy in patients with Colorectal Cancer from stage II to IV

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* Determine the response rate in patients with Colorectal Cancer treated with Cetuximab and Radiation Therapy Vs Surgery before or after Radiation Therapy.

Secondary:

* To determine the progression-free survival and overall survival of patients treated with these regimens.
* Compare the treatment compliance of patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is an Open-label, Controlled, Multicenter study. Patients will be assigned into two different Arms.

Arm I: Patients will receive Cetuximab and Radiation Therapy. Patients will receive a dose of Cetuximab through Intravenous (IV). The initial dose is 400 mg/m2 administered as a 120-minute intravenous infusion (maximum infusion rate 10 mg/min) and weekly dose is 250 mg/m2 infused over 60 minutes (maximum infusion rate 10 mg/min) until disease progression or unacceptable toxicity. Radiation treatment for Colorectal Cancer are Intensity Modulated Radiation Therapy (IMRT). IMRT delivers radiation directly to the tumor and modulates the intensity of the radiation with laser accuracy.

Arm II: Patients will undergo surgery before or after Radiation Therapy. Colorectal Cancer Surgery are Colon resection (Colectomy), Rectum resection (Proctectomy), Colostomy, and Radiofrequency ablation. Radiation treatment for Colorectal Cancer are Intensity Modulated Radiation Therapy (IMRT). IMRT delivers radiation directly to the tumor and modulates the intensity of the radiation with laser accuracy.

PROJECTED ACCRUAL: Approximately 450 patients will be accrued for this study within 18 to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II- IV Colorectal Cancer
* Patients must be 40 years and older
* Patients may be of any race and either gender
* Signed Informed Consent

Patient characteristics:

* Age: 40 years and older
* Sex: Both
* Performance status: Not specified
* Life expectancy: Not specified

Hematopoietic:

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* No history of significant bleeding events within the past 6 months

Hepatic:

* Bilirubin ≤ 1.5 mg/dL
* Albumin ≥ 2.5 g/dL

Renal:

* Creatinine ≤ 1.5 times upper limit of normal
* Protein < 1+ by urinalysis
* Protein < 1 g by 24-hour urine collection

Cardiovascular:

* No conduction defect in heart
* No congestive heart failure
* No myocardial infarction within last 6 months
* No cerebrovascular accident
* No uncontrolled hypertension
* No clinically significant peripheral artery disease

Pulmonary:

* No pulmonary embolism
* No interstitial pneumonia
* No extensive or symptomatic interstitial fibrosis of the lung

Neurologic:

* No uncontrolled seizure disorder
* No active neurological disease

Other:

* Not pregnant or nursing
* Negative pregnancy test

Exclusion Criteria:

* Age below 40 years
* Brain or nervous system metastases
* Any current mental illness
* Hemoglobin is less than 9.0 g/dl
* CBC results are below normal range
* Patients with Hepatitis B or C or who are HIV positive
* Pregnant or nursing patients are not eligible for entry into the study
* Hepatic abnormality AST/ALT > 4 folds

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response rate | 4 year

SECONDARY OUTCOMES:
Tolerability | 4 years
Progression free survival | 4 years
Overall survival | 4 Years
Quality of life | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Grewal, MD, Study Chair — American Scitech International- eCRO; Prem A Nandiwada, MD, Principal Investigator — Raritan Bay Medical Center; Sarat Babu, MD, Study Director — St. Peter's Hospital; S N Agrawal, MD, Principal Investigator — JLR Hospital in India
Locations (1):
- Practicing Physician in New Jersey, Englishtown, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.imclone.com
- See also: Related Info — http://www.bristolmyers.com